CLINICAL TRIAL: NCT00306319
Title: Pharmacokinetic Interaction Study of Rifampicin, Isoniazid and Moxifloxacin in Tuberculosis Patients in Bandung, Indonesia
Brief Title: Pharmacokinetic Interaction Study in Indonesian Tuberculosis Patients Indonesia
Status: Completed | Phase: Phase 2 | Type: Interventional
Sponsor: Radboud University Medical Center (Other)
Allocation: Non-Randomized | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: UMCN-AKF 05.02; Primo study
Record Dates: First submitted 2006-03-22; First posted 2006-03-23 (Estimated); Last update posted 2020-11-12 (Actual); Status verified 2020-11

CONDITIONS: Tuberculosis
Keywords: Tuberculosis
MeSH Terms: conditions — Tuberculosis | interventions — Moxifloxacin

INTERVENTIONS:
Drug: moxifloxacin

SUMMARY:
Pharmacokinetic study in TB patients to determine the effect of rifampicin on the pharmacokinetic profile of moxifloxacin.

DETAILED DESCRIPTION:
Tuberculosis is an infectious disease that still causes many victims in the developing world, especially in Indonesia. Rifampicin, isoniazid and ethambutol are the cornerstone of the current treatment. The disadvantage of the current treatment is the long, six-months, duration of the treatment. This long duration contributes to suboptimal adherence to the TB drugs.Thus, there is a very urgent need to evaluate drugs that may help shortening TB treatment. The fluoroquinolone moxifloxacin has shown early bactericidal activity (EBA) in patients with pulmonary TB, and has shown rapid and reliable sterilization. Rifampicin is a strong inducer of the CYP enzymes, but it also induces phase II metabolism. As moxifloxacin is metabolized by phase II metabolism, rifampicin could cause a decrease in the plasma concentrations of moxifloxacin. Therefore, a pharmacokinetic interaction study is warranted.

ELIGIBILITY:
Inclusion Criteria:

* Indonesian AFB negative tuberculosis patients who are in the last two months of the continuation phase of their six-month-antituberculosis treatment.
* Subject is 18-55 years of age at the day of the first dosing of study medication.
* Subject has a normal ECG
* Subjects bodyweight is >35kg
* Use of rifampicin and isoniazid

Exclusion Criteria:

* Pregnant or lactating
* History or condition that might interfere with drug absorption, distribution, metabolism or excretion, including ileus, gastric paresis, liver and renal dysfunction, diabetes mellitus.
* Presence of contraindications for moxifloxacin or use of drugs that are known to interact with moxifloxacin.
* Subject is not able and/or not willing to sign the informed consent form.

Ages: 18 Years to 55 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult
Enrollment: 23
Dates: Start 2006-01; Primary Completion 2006-05 (Actual); Study Completion 2006-05 (Actual)

PRIMARY OUTCOMES:
Pharmacokinetic (24 hrs) curves will be drawn
at day 5 in period I and period II.

CONTACTS AND LOCATIONS:
Overall Officials: R. Aarnoutse, PharmD PhD, Principal Investigator — Radboud University (RUNMC)
Locations (1):
- Rumah Sakit Hasan Sadikin (RSHS), Bandung, Indonesia

REFERENCES:
- [Result] Nijland HM, Ruslami R, Suroto AJ, Burger DM, Alisjahbana B, van Crevel R, Aarnoutse RE. Rifampicin reduces plasma concentrations of moxifloxacin in patients with tuberculosis. Clin Infect Dis. 2007 Oct 15;45(8):1001-7. doi: 10.1086/521894. Epub 2007 Sep 4. PMID 17879915